CLINICAL TRIAL: NCT05765474
Title: Motor Learning for Individuals With Upper Limb Hemiparesis After Stroke
Brief Title: Motor Learning for Upper Limb Hemiparesis After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Dawn Nilsen, Professor of Rehabilitation and Regenerative Medicine, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: AAAU1704
Record Dates: First submitted 2023-03-01; First posted 2023-03-13 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-08

CONDITIONS: Stroke; Hemiparesis
Keywords: Stroke; Hemiparesis; Rehabilitation; Motor Learning
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Research participants will be blinded to the overall purpose of the study and will not be informed of the difference between the groups. They will be debriefed after the completion of all study procedures in accordance with IRB policies. Outcomes assessors will be blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Training with Practice Variable (Experimental): All participants will practice a motor task (the Scooping Task) for 2 consecutive days. Each day of training, participants will complete 50 trials (10 blocks of 5 trials each) with their more affected arm and 20 trials (10 blocks of 2 trials each) with their less affected arm. One trial of the task will involve using a spoon to scoop beans, one at a time, from one cup to another while seated at a table. Participants will be asked to complete as many scoops as possible from the cup closest to them to the cup farthest from them within 30 seconds in an anterior-posterior direction. One successful repetition occurs when at least one bean is transferred. The number of successful repetitions within a 30 second trial is then counted. Training for the experimental group will include the practice variable of interest.
  Interventions: Behavioral: Practice Variable
- Training without Practice Variable (Other): All participants will practice a motor task (the Scooping Task) for 2 consecutive days. Each day of training, participants will complete 50 trials (10 blocks of 5 trials each) with their more affected arm and 20 trials (10 blocks of 2 trials each) with their less affected arm. One trial of the task will involve using a spoon to scoop beans, one at a time, from one cup to another while seated at a table. Participants will be asked to complete as many scoops as possible from the cup closest to them to the cup farthest from them within 30 seconds in an anterior-posterior direction. One successful repetition occurs when at least one bean is transferred. The number of successful repetitions within a 30 second trial is then counted. Training for the control group will not include the practice variable of interest.
  Interventions: Behavioral: No Practice Variable

INTERVENTIONS:
Behavioral: Practice Variable — This group receives the practice variable. The practice variable being studied will not be disclosed until completion of testing procedures.
  Arms: Training with Practice Variable
Behavioral: No Practice Variable — This group does not receive the practice variable. The practice variable being studied will not be disclosed until completion of testing procedures.
  Arms: Training without Practice Variable

SUMMARY:
The purpose of this research is to learn about practice conditions that may benefit stroke survivors when learning to use their more affected arm to perform a task. Participants will be randomized into two groups. Experimental and control groups will differ by one practice variable that will not be disclosed until completion of testing procedures. Participants will practice a motor task using both their more and less affected arms for two consecutive days. A Pre-Test will be administered on Day 1 before the training begins. Immediate Transfer of Learning will be administered on Day 2 after the completion of training. Delayed (24-hour) Retention and Transfer Tests will be administered on Day 3.

DETAILED DESCRIPTION:
Stroke involves loss of blood flow to the brain and can cause impaired upper limb motor function, resulting in long term disability. Targeted motor learning interventions can improve skill acquisition and functional upper limb use after stroke. For example, repetitive practice of a motor task has been shown to improve motor learning outcomes. However, more research is currently needed to identify important active ingredients in complex motor learning interventions and determine the most effective approaches for improving upper limb recovery after stroke. The purpose of this study is to investigate the impact of a specific practice variable on motor learning for individuals with upper limb hemiparesis after stroke. This research will inform the development of future stroke rehabilitation interventions aimed at improving skill acquisition and motor learning.

ELIGIBILITY:
Inclusion Criteria:

* At least 6 months following stroke (ischemic or hemorrhagic)
* Upper limb weakness resulting from the stroke
* Able to follow 2-step commands
* Box and Block test score of 3-60
* Intact proprioception at the index finger of the weaker arm
* English speaking

Exclusion Criteria:

* Severe neglect (Score of 2 on extinction and inattention items of NIHSS)
* Arm pain that limits movement or loss of functional range of movement (contracture)
* Unable to give informed consent
* Received Botox within the past 3-months

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-03-22 (Actual); Primary Completion 2024-02-16 (Actual); Study Completion 2024-02-16 (Actual)

PRIMARY OUTCOMES:
24-Hour Retention Test: Number of completed scoops (more affected arm) | Day 3
  This is a 24-hour Retention Test of the trained motor task (the Scooping Task) that the participant practiced for 2 days. The participant is asked to use a spoon to scoop beans from one cup to another in an anterior-posterior direction, away from their body, for 30 seconds. One completed scoop occurs when at least one bean is transferred to the second cup. The score is the number of completed scoops that occur within 30 seconds. The participant will complete two blocks of five trials (30 seconds each). The number of completed scoops will be averaged across blocks of trials.

SECONDARY OUTCOMES:
Immediate Transfer Test: Number of transported cubes (more affected arm) | Day 2
  This is an Immediate Transfer Test that will be administered on Day 2 following completion of training on the Scooping Task. The participant is asked to transport cubes in an anterior-posterior direction away from their body, using the Box and Block Test apparatus, for 30 seconds. The score is the number of cubes that are transported within 30 seconds. The participant will complete two blocks of five trials (30 seconds each). The number of transported cubes will be averaged across blocks of trials.
24-Hour Transfer Test: Number of transported cubes (more affected arm) | Day 3
  This is a 24-Hour Transfer Test that will be administered on Day 3. The participant is asked to transport cubes in an anterior-posterior direction away from their body, using the Box and Block Test apparatus, for 30 seconds. The score is the number of cubes that are transported within 30 seconds. The participant will complete two blocks of five trials (30 seconds each). The number of transported cubes will be averaged across blocks of trials.
Self-Efficacy Rating for Scooping Task | Day 2
  After completing training on Day 2, the participant will be asked to rate their confidence in achieving various scores on the trained motor task (the Scooping Task). Self-Efficacy will be rated using a 10 point scale (0 = Not confident at all; 10 = Very confident) with higher scores indicating a better outcomes. Scores will be calculated by averaging Self-Efficacy ratings.
Rating of Mood | Day 2
  After completing training on Day 2, participants will be asked to rate their mood using the valence subscale of the Self-Assessment Manikin, which is a non-verbal assessment of affect that has five pictures of smiling, neutral, and frowning faces. The participant rates their mood using a 9 point scale based on the pictures (1 = More positive affect; 9 = Less positive affect) with lower scores indicating a better outcome.
Interest/Enjoyment Subscale of the Intrinsic Motivation Inventory | Day 2
  After completing training on Day 2, the participant will complete items from the interest/enjoyment subscale of the Intrinsic Motivation Inventory. This is an assessment of participant's subjective experience of the Scooping Task. Participants will rate each statement according to how true it is for them, using a 7 point scale (1 = Not true at all; 7 = Very true). Higher scores indicate greater interest/enjoyment when practicing the task (better outcome). Scores are calculated by averaging the item scores of the subscale.
Perceived Competence Subscale of the Intrinsic Motivation Inventory | Day 2
  After completing training on Day 2, the participant will complete items from the perceived competence subscale of the Intrinsic Motivation Inventory. This is an assessment of participant's subjective experience of the Scooping Task. Participants will rate each statement according to how true it is for them, using a 7 point scale (1 = Not true at all; 7 = Very true). Higher scores indicate greater perceived competence when practicing the task (better outcome). Scores are calculated by averaging the item scores of the subscale.
Perceived Choice Subscale of the Intrinsic Motivation Inventory | Day 2
  After completing training on Day 2, the participant will complete items from the perceived choice subscale of the Intrinsic Motivation Inventory. This is an assessment of participant's subjective experience of the Scooping Task. Participants will rate each statement according to how true it is for them, using a 7 point scale (1 = Not true at all; 7 = Very true). Higher scores indicate greater perceived choice when practicing the task (better outcome). Scores are calculated by averaging the item scores of the subscale.
Value Subscale of the Intrinsic Motivation Inventory | Day 2
  After completing training on Day 2, the participant will complete items from the value subscale of the Intrinsic Motivation Inventory. This is an assessment of participant's subjective experience of the Scooping Task. Participants will rate each statement according to how true it is for them, using a 7 point scale (1 = Not true at all; 7 = Very true). Higher scores indicate greater value associated with the task (better outcome). Scores are calculated by averaging the item scores of the subscale.
Effort Subscale of the Intrinsic Motivation Inventory | Day 2
  After completing training on Day 2, the participant will complete items from the effort subscale of the Intrinsic Motivation Inventory. This is an assessment of participant's subjective experience of the Scooping Task. Participants will rate each statement according to how true it is for them, using a 7 point scale (1 = Not true at all; 7 = Very true). Higher scores indicate greater effort associated with the task (better outcome). Scores are calculated by averaging the item scores of the subscale.
Pressure/Tension Subscale of the Intrinsic Motivation Inventory | Day 2
  After completing training on Day 2, the participant will complete items from the pressure/tension subscale of the Intrinsic Motivation Inventory. This is an assessment of participant's subjective experience of the Scooping Task. Participants will rate each statement according to how true it is for them, using a 7 point scale (1 = Not true at all; 7 = Very true). Higher scores indicate greater pressure/tension when practicing the task (worse outcome). Scores are calculated by averaging the item scores of the subscale.

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Nilsen, EdD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States